CLINICAL TRIAL: NCT05804279
Title: Pharmacokinetics and Safety of BPDO-1603 or BPDO-16031 and BPDO-16033 Administration in Healthy Adults. Randomized, Open-label, Single-dose, Cross-over, Phase 1 Study
Brief Title: Pharmacokinetics of BPDO-1603 or BPDO-16031 and BPDO-16033 Administration in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-007-05
Record Dates: First submitted 2023-03-15; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Alzheimer's disease, Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPDO-1603 (Experimental): 1 tablet contains memantine 20mg/donepezil 10mg
  Interventions: Drug: BPDO-1603
- BPDO-16031,BPDO-16033 (Active Comparator): 1 tablet memantine 20mg and 1 tablet donepezil 10mg
  Interventions: Drug: BPDO-1603

INTERVENTIONS:
Drug: BPDO-1603 — donepezil/mematine

SUMMARY:
Pharmacokinetics and safety of BPDO-1603 or BPDO-16031 and BPDO-16033 administration in healthy adults. Randomized, open-label, single-dose, cross-over, Phase 1 study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 or older and 55 or less at the time of screening tests
2. Men weigh 55 kg or more and women weigh 50 kg or more
3. Those with a body mass index of 18.5 kg/m2 or more and less than 27.0 kg/m2

Exclusion Criteria:

1. Clinically significant active chronic diseases, hepatometer (severe liver disorder, etc.), kidney (severe kidney disorder, etc.), and nervous system (hepatorespiratory tract patients). Parkinson's disease, immune system, respiratory system (asthenia, obstructive pulmonary disease, etc.), urinary system, digestive system (digestive ulcer, etc.), endocrine system, blood/tumor, cardiovascular system (cardiac infarction, heart failure, uncontrolled hypertension, atrioventricular junction disorder, etc.), or have a history.
2. A person who has a serious urinary tract infection due to renal tubular acidosis, etc. or has a history of history
3. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Cmax of memantine and donpezil | from baseline to day 10
  pharmacokinetic properties

SECONDARY OUTCOMES:
AUClast of memantine and donpezil | from baseline to day 10
  pharmacokinetic properties

CONTACTS AND LOCATIONS:
Locations (1):
- Hyundaipharm, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided